CLINICAL TRIAL: NCT04540458
Title: Effect of 3D Ultrasounds and 3D Printed Models on Maternal and Paternal Fetal Attachment and Anxiety and Depression
Brief Title: 3D Maternal Fetal Bonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1052761
Record Dates: First submitted 2020-03-16; First posted 2020-09-07 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Maternal-Fetal Relations; Paternal Behavior; Maternal Behavior

STUDY DESIGN:
Intervention Model Description: 3D ultrasound and picture of ultrasound or 3D ultrasound and printed model of fetal face
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed model (Other): Mother or Mother/Father is given 3D printed model of fetus' face
  Interventions: Other: 3D printed model
- Placebo (Other): Mother or Mother/Father is given printed picture of 3D ultrasound of fetus
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 3D printed model — Mother or Mother/Father is given 3D printed model of fetus' face
  Arms: 3D printed model
Other: Placebo — Mother or Mother/Father is given a picture of 3D ultrasound of fetus
  Arms: Placebo

SUMMARY:
To determine whether 3D models of fetus' face created from 3D ultrasound will increase maternal and paternal attachment, lower stress, anxiety and depression and have improved life-style choices during pregnancy. Half of participants will receive 3D model and half will receive a picture of 3D ultrasound of their baby.

ELIGIBILITY:
Inclusion Criteria:

* Age - Female 19-45 years of age; Male > 19 years of age
* Currently pregnant (< 32 weeks gestation)
* Have normal 20-week ultrasound

Exclusion Criteria:

* Having received more than 3 ultrasounds prior to study
* Medical need for additional ultrasounds
* Multiple fetuses
* > 31 weeks gestation

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Maternal Antenatal Attachment Scale (MAAS) | 5 minutes
  The MAAS is a 19 item questionnaire measuring maternal-fetal attachment. Each item has five answer choices scored from 1 low attachment to 5 high attachment such that the total score ranges from 19 to 95. The measure also includes two subscales: (1) Quality of Attachment has 10 items with a range of 10-50 and measures the quality of the mother's attachment to her fetus. (2) Time measures the time spent in attachment mode (or intensity of preoccupation) and consists of 8 items for a range of 8 to 40. (for clarity one item included in the total score is not included in either subscale.)
Paternal Antenatal Attachment Scale (PAAS) | 5 minutes
  The PAAS is a 16 item questionnaire measuring paternal-fetal attachment. Each item has five answer choices scored from 1 low attachment to 5 high attachment such that the total score ranges from 19 to 95. The measure also includes two subscales: (1) Quality of Attachment has 10 items with a range of 10-50 and measures the quality of the mother's attachment to her fetus. (2) Time measures the time spent in attachment mode (or intensity of preoccupation) and consists of 8 items for a range of 8 to 40. (for clarity one item included in the total score is not included in either subscale.)
Maternal anxiety | 3 minutes
  7-question Generalized Anxiety Disorder questionnaire (GAD-7) will be administered
Paternal depression | 3 minutes
  9-question Patient Health Questionnaire (PHQ-9) will be administered
Maternal depression | 3 minutes
  9-question Patient Health Questionnaire (PHQ-9) will be administered
Paternal anxiety | 3 minutes
  7-question Generalized Anxiety Disorder questionnaire (GAD-7) will be administered
Maternal stress | 3 minutes
  11-question Pregnancy-Related Anxiety Questionnaire-Revised (PRAQ-R2) will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: John Cote, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No